CLINICAL TRIAL: NCT00329979
Title: Silent Cerebral Infarction After Heart Catheterization: A Randomized Comparison of Radial and Femoral Arterial Access.
Brief Title: Femoral vs Radial Approach and MRI Evaluation of Strokes
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Patrick MICHEL, research and strategy manager, University hospital, Caen
Other Study IDs: 2006-18; No additional Ids
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; radial; femoral; vascular access site; embolism; cerebral; MRI; stroke
MeSH Terms: conditions — Aortic Valve Stenosis; Embolism; Stroke

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Radial access
  Interventions: Behavioral: vascular access site
- 2: Femoral access
  Interventions: Behavioral: vascular access site

INTERVENTIONS:
Behavioral: vascular access site — Randomized vascular access site

SUMMARY:
Symptomatic cerebral infarction following cardiac catheterization is rare but silent brain injury could occur at an unexpectedly high rate. One study has found that up to 22% of patients with severe aortic stenosis who have undergone retrograde catheterization of the valve can be identified as having new ischemic lesions as detected by diffusion-weighted (DW) magnetic resonance imaging (MRI). During cardiac catheterization, cerebral microembolism as detected by TCD has frequently been observed, but whether it is clinically relevant remains unknown . However, recent studies have suggested that some of these microemboli could be responsible for acute brain injury, as documented by DW MRI.

Indeed the high sensitivity of DW MRI suggests that this technique could allow an improved estimate of cerebral ischemic events associated with cardiovascular-catheter procedures. We therefore decided to perform DW MRI before and after cardiac catheterization to prospectively assess both clinically silent and apparent cerebral embolisms for the first time in a multicenter trial. Furthermore, a randomization between radial and femoral access will allow assessment of risk of silent brain injury associated with the different vascular access sites.

ELIGIBILITY:
Inclusion Criteria:

* Patient with significant aortic valve stenosis before planned surgery.

Exclusion Criteria:

* Contraindication to MRI or inability to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Hamon, MD, Study Chair — CHU CAEN; Martial Hamon, MD, Principal Investigator — CHU CAEN
Locations (1):
- CHU Caen, cardiology department, Caen, France